CLINICAL TRIAL: NCT04214587
Title: Biological Investigation of Explanted Endobronchial Lung Valves Study - Investigation of the Mechanism of Action of Tissue-device Interactions
Brief Title: Biological Investigation of Explanted Endobronchial Lung Valves Study
Acronym: Bio-EXCEL
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, Prof. dr. D.J. Slebos MD, PhD, Principle Investigator, University Medical Center Groningen
Other Study IDs: Bio-EXCEL
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Emphysema or COPD
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive | interventions — Histocompatibility Testing; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — epithial brushings blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- baseline assessment group: n=150 patiënts for baseline assessment
  Interventions: Diagnostic Test: tissue and blood sampling
- clinical need for reintervention group: n=20-30 patiënts for re-bronchoscopy
  Interventions: Diagnostic Test: tissue and blood sampling
- clinical stable controls: n=20 stable treated control patiënts
  Interventions: Diagnostic Test: tissue and blood sampling

INTERVENTIONS:
Diagnostic Test: tissue and blood sampling — only diagnostics will be peformed

SUMMARY:
Rationale:

COPD is a severe, often progressive and currently incurable lung disease which affects both the upper airways (chronic bronchitis) as well as the lower airways (emphysema). In advanced stages of the disease air-trapping severely reduces the ability to breathe and subsequently the quality of life. A highly effective treatment for restoring lung mechanical functionality of these patients is the introduction of bronchoscopic lung volume reduction (BLVR), e.g. implanting small silicone/nitinol valves (EBV) inside the airways to reduce air-trapping. Although successfully investigated in a selected group of severe COPD patients, the effectiveness of the treatment can sometimes be short-lived due to fibrotic and granulation responses and tissue-material interactions.

Objective:

The main objective of this study is to study and understand the underlying biological principles of granulation and fibrotic responses limiting the effectiveness and longevity of BELVR treatment with EBVs, this to investigate the mechanism of action of tissue-device interactions.

ELIGIBILITY:
Inclusion Criteria:

* Elidgible for EBV treatment

Exclusion Criteria:

* Anticoagulation which cannot be stopped prior to the procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severe emphysema patients routinely scheduled for bronchoscopic lung volume reduction with one-way endobronchial valves
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2027-03-02 (Estimated); Study Completion 2027-03-02 (Estimated)

PRIMARY OUTCOMES:
the % of the 150 patients that will develop a need for rebronchoscopy after 18 months | 18 months
  frequency

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD PhD, Principal Investigator — UMC-Groningen/NL
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The UMC-Groningen/NL Bronchoscopic Intervention Center website — http://www.bicumcg.nl